CLINICAL TRIAL: NCT04581343
Title: A Phase 1B Study to Determine the Safety and Tolerability and Confirm the Dose of Canakinumab and Spartalizumab in Combination With Nab-paclitaxel and Gemcitabine for Patients With Metastatic Pancreatic Cancer
Brief Title: A Phase 1B Study of Canakinumab, Spartalizumab, Nab-paclitaxel, and Gemcitabine in Metastatic Pancreatic Cancer (PC) Patients
Acronym: PanCAN-SR1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pancreatic Cancer Action Network (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PanCAN-SR1
Record Dates: First submitted 2020-09-14; First posted 2020-10-09 (Actual); Results first posted 2025-04-08 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — canakinumab; spartalizumab; 130-nm albumin-bound paclitaxel; Gemcitabine; Albumin-Bound Paclitaxel

STUDY DESIGN:
Intervention Model Description: A Phase 1B study enrolling 10 patients to find 6 evaluable patients starting at a maximum dose. If Dose Limiting Toxicities are noted a lower dose may be evaluated to determine the recommended Phase II dose level.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Canakinumab, spartalizumab, nab-paclitaxel and gemcitabine (Experimental): Spartalizumab (PDR001),IV infusion, 400 mg, D1 of each 28-day cycle; Canakinumab (ACZ885), s.c. injection, 250 mg, Day 1 of each 28- day cycle; Gemcitabine, IV Infusion, 1000 mg/m2, Days 1, 8, 15 of each 28-day cycle; Nab-paclitaxel, IV Infusion, 125 mg/m2, Days 1, 8, 15 of each 28-day cycle.
  Interventions: Drug: Canakinumab injection; spartalizumab, nab-paclitaxel, gemcitabine

INTERVENTIONS:
Drug: Canakinumab injection; spartalizumab, nab-paclitaxel, gemcitabine — Canakinumab 250 mg s.c. injection; Spartalizumab 400 mg IV infusion, nab-paclitaxel 125 mg/m2 IV infusion, gemcitabine 1000 mg/m2 IV infusion
  Other Names: Ilaris; Abraxane

SUMMARY:
This study combines canakinumab (ACZ885), a high-affinity human anti-interleukin-1β (IL-1β) monoclonal antibody (mAb), and spartalizumab (PDR001), a mAb directed against human Programmed Death-1 (PD-1), with the chemotherapy combination of gemcitabine and nab-paclitaxel. This study will confirm for this 4-drug combination the tolerable doses, the acceptable safety profile, and the dose to be used for a Phase II combination treatment regimen.

DETAILED DESCRIPTION:
This is an open-label multi-center phase Ib study to confirm the recommended phase II/III dose of canakinumab and spartalizumab in combination with nab-paclitaxel and gemcitabine.

The study will recruit patients with metastatic pancreatic adenocarcinoma treated in the first line setting. The starting dose level of canakinumab explored will be 250 mg Q4W ("starting dose level"). In case of unacceptable toxicity of the starting dose level of canakinumab, the dose of canakinumab will be de-escalated to the "-1 dose level" administered as 250 mg Q8W, while other components of the combination stay at the same dose as the starting dose level.

Patients will be observed for dose limiting toxicities (DLTs) for a minimum duration of 56 days (8 weeks). To achieve study objectives and to ensure the adequate number of DLT evaluable patients, the study will recruit approximately ten patients to have at least 6 evaluable patients per dose level of canakinumab. Additional approximately ten patients (to have at least 6 additional evaluable patients) may be enrolled at lower dose level in case a dose de-escalation is necessary.

Dose confirmation will be guided by an adaptive Bayesian logistic regression model (BLRM) based on any DLTs observed for two cycles of treatment (i.e. 56 days, or 8 weeks). The adaptive BLRM will be guided by the Escalation with Overdose Control (EWOC) principle to control the probability of DLT in future patients on the study. BLRM is a well-established and widely used method to estimate the recommended dose for expansion (RDE) or maximal tolerable dose (MTD) in clinical trials in patients with cancer with small sample size. The use of Bayesian response adaptive models for small datasets has been endorsed by academic publications (Babb et al. 1998, Neuenschwander et al. 2008, Neuenschwander et al. 2010, Natanegara et al. 2014), by the European Medicines Agency (Guideline on Clinical Trials in Small Populations, 2007) and it constitutes an important aspect of the FDA's Critical Path Initiative (Clinical Path White Paper, FDA, 2004). The Bayesian analysis incorporates prior toxicity data of single agent and drugs combinations together with the currently available data to predict the probability of DLT and excessive toxicity of a dose level of interest.

The Bayesian method is be based on a Meta-Analytical-Combined (MAC) approach (Spiegelhalter 2004, Neuenschwander 2016) to combine all historical and concurrent data. Prior toxicity information included in the BLRM model was obtained from three studies with canakinumab as a single agent and combination of canakinumab and spartalizumab (PDR001X2101, ACZ885I2202, PRD001X2103) and from a phase I/II study of nab-paclitaxel + gemcitabine (Von Hoff D, et.al., 2011). Simulation was used to illustrate the recommendation from BLRM under a set of hypothetical scenarios with assumed number of evaluable patients and DLTs.

The decisions on a recommended dose will be made by the Investigators and the Sponsor in a Safety Review meeting when at least 6 DLT evaluable patients per dose level will be observed for DLTs for a minimum duration of 56 days (8 weeks). Safety review will be based upon the review of all relevant data available including treatment tolerability and safety information together with the BLRM summaries of DLT probability, PK, PD, and preliminary activity information (if available) at the time of the meeting.

Patients will be treated until disease progression per RECIST 1.1, unacceptable toxicity, or until the patient or treating physician decides to stop treatment.

Pharmacokinetic (PK) and immunogenicity (IG) samples will be collected at specific time points throughout treatment. Each treatment cycle is 4 weeks. All patients must be followed for safety up to 150 days after the last dose of spartalizumab or canakinumab, or 30 days after the last dose of the combination chemotherapy, whichever the later. After the end of safety follow-up, patients will be followed for disease progression if discontinuation of treatment is due to reason other than progression, and for survival (via telephone call or onsite visit if a patient happens to be visiting the site) until the end of study The study completion is defined as when the last patient has completed the study treatment, safety follow up, and completed survival follow up period up to 1 year from first treatment, whichever is later or in the event of an early study termination decision, the date of that decision.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years at the time of informed consent
* Histologically or cytologically confirmed pancreatic ductal adenocarcinoma (PDAC) (determined by a local laboratory) with metastatic spread of disease (adenosquamous is also allowed).
* Patients must have not received previous anti-cancer therapy for the treatment of metastatic pancreatic ductal adenocarcinoma.
* Patients who received previous neo-/adjuvant systemic therapy for non-metastatic PDAC ≥12 months from the last treatment to study enrollment date are allowed unless this therapy included immunotherapy and/or IL-1 inhibitors.
* Radiographically measurable disease of at least one site by computed tomography (CT) scan (or magnetic resonance imaging, if allergic to CT contrast media) as defined by Response Evaluation Criteria In Solid Tumors (RECIST 1.1). Primary lesion is allowed as long as it is measurable (per RECIST 1.1) and has not been previously irradiated. Imaging results must be obtained within the 28-day screening window.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Adequate organ function (laboratory results must be obtained within the 28-day screening window)

  * Absolute neutrophil count > 1500/mm3
  * Hemoglobin > 9 g/dL
  * Platelets > 100,000/mm3
  * Serum creatinine < 1.5 x upper limit normal (ULN), or calculated creatinine clearance > 60 mL/min (Cockcroft Gault)
  * Albumin > 3.0 g/dL
  * Aspartate aminotransferase (AST) serum glutamic oxaloacetic transaminase (SGOT) and/or alanine aminotransferase (ALT) serum glutamic pyruvic transaminase (SGPT) < 3.0 x ULN (< 5 x ULN in presence of liver metastasis).

In patients with elevated ALT or AST, the values must be stable for at least 2 weeks and with no evidence of biliary obstruction on imaging

* Total bilirubin ≤ 1.5 X ULN
* INR ≤ 1.5 x ULN

  * Consent to provide protocol-mandated tissue and blood samples for diagnostic, PK, and research purposes
  * Able to adhere to study visit schedule and other protocol requirements

Exclusion Criteria:

* Diagnosis of pancreatic neuroendocrine carcinoma or pancreatic acinar cell carcinoma
* Previous immunotherapy (e.g. anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways).
* Known microsatellite instability-high (MSI-H) or mismatch repair-deficient pancreatic cancer
* Prior treatment with canakinumab or drugs of a similar mechanism of action (IL-1 inhibitor).
* History of known hypersensitivity to any of the drugs used in this study or any of their excipients, or patient has contraindication to any of the study drugs as outlined in the local prescribing information (e.g. United States Prescribing Information [USPI])
* Active autoimmune disease that has required systemic treatment in the past 2 years prior to enrollment i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs. Control of the disorder with replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is permitted.
* Patient with suspected or proven immunocompromised state or infections, including:

  * Evidence of active or latent tuberculosis (TB) as determined by locally approved screening methods. If the results of the screening per local treatment guidelines or clinical practice require treatment, then the patient is not eligible.
  * Chronic or active hepatitis B or C
  * Known history of testing positive for Human Immunodeficiency Virus (HIV) infections.
  * Any other medical condition (such as active infection, treated or untreated), which in the opinion of the investigator places the patient at an unacceptable risk for participation in immunomodulatory therapy.

Note: Patients with localized condition unlikely to lead to a systemic infection e.g. chronic nail fungal infection are eligible.

* Allogeneic bone marrow or solid organ transplant
* Treatment with any immune modulating agent in doses with systemic effects e.g.:

  * Systemic treatment with prednisone > 10 mg (or equivalent) for >14 days within 4 weeks prior to the first dose of study treatment.
  * Equivalent dose of methotrexate > 15 mg weekly
  * Patient receiving any biologic drugs targeting the immune system (for example, TNF blockers, anakinra, rituximab, abatacept, or tocilizumab).
  * Note: Daily glucocorticoid-replacement for conditions such as adrenal or pituitary insufficiency is allowed.
  * Note: Topical, inhaled, or local steroid use in doses that are not considered to cause systemic effects are permitted (based on investigator's discretion and consultation with the Medical Monitor if needed).
* Patient has concurrent malignancy other than the disease under investigation, with exception of malignancy that was treated curatively and has not recurred within 2 years prior to the date of screening. Fully resected basal or squamous cell skin cancers, and any carcinoma in situ are eligible.
* Uncontrolled or severe cardiac disease (history of unstable angina, myocardial infarction, coronary stenting, or bypass surgery within the prior 6 months), symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia [including atrial flutter/fibrillation], requirement for inotropic support or use of devices for cardiac conditions [pacemakers/defibrillators]), uncontrolled hypertension defined by a systolic blood pressure =>160 mg and/or diastolic blood pressure =>100 mg Hg
* Pre-existing peripheral neuropathy > Grade 1 (CTCAE V 5.0)
* Receipt of live vaccines within 3 months prior to the first dose of study treatment or while on active treatment within the trial (examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid (oral vaccine). Seasonal influenza vaccines for injection are generally killed virus vaccines and are permitted. However, intranasal influenza vaccines (e.g. Flu-mist) are live attenuated vaccines and are not permitted.
* Patient has had major surgery within 14 days prior to enrollment
* Patient has symptomatic brain metastases, or brain metastases that require directed therapy (such as focal radiotherapy or surgery). Patients with treated brain metastases have to be neurologically stable and not using systemic steroids for at least 4 weeks prior to the study drug administration.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are willing to use highly effective methods of contraception during treatment with study drugs (canakinumab, spartalizumab, gemcitabine and nab-paclitaxel).
* Highly effective contraception methods are required while on treatment and for 150 days after stopping spartalizumab. No contraception is required after treatment with canakinumab is stopped. Contraception use after chemotherapy is stopped should be followed per the local drug label requirements.

Highly effective contraception methods include:

* Total abstinence (when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (i.e., calendar, ovulation, symptothermal, postovulation methods) and withdrawal are not acceptable methods of contraception
* Female sterilization (have had bilateral surgical oophorectomy (with or without hysterectomy), total hysterectomy or bilateral tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
* Male sterilization (at least 6 months prior to screening). The vasectomized male partner should be the sole partner for that patient.
* Use of oral, injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS) or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment.

Note: Women of non-childbearing potential is defined as women who are physiologically and/or anatomically incapable of becoming pregnant, as now further described:

* They are post-menopausal as evidenced by 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (i.e., age appropriate history of vasomotor symptoms).
* They have had bilateral surgical oophorectomy (with or without hysterectomy), total hysterectomy or bilateral tubal ligation at least six weeks prior. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of childbearing potential.

Note: Sexually active male patients and their partners who are women of childbearing potential should follow the contraception recommendations and any other precautionary measures as required by the local prescribing information for the standard of care (SOC) anti-cancer.

* Any significant medical condition, laboratory abnormality or psychiatric condition that would constitute unacceptable safety risks to the patients, contraindicate patient participation in the clinical study, limit the patient's ability to comply with study requirements, or compromise patient's compliance with the protocol and all requirements of the study as stated in the Informed Consent Form. Significant medical conditions include but are not limited to known history or current interstitial lung disease or non-infectious pneumonitis, medical history or current diagnosis of myocarditis, chronic active hepatitis, liver cirrhosis or any other significant liver disease with moderate to severe hepatic impairment (Child-Pugh B or C), serious non-healing wound/ulcer/bone fracture, uncompensated/symptomatic hypothyroidism, or requirement for hemodialysis or peritoneal dialysis.
* Unwillingness or unable to comply with all requirement of the study as stated in the Informed Consent Form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2023-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Berkenbilt, Study Director — Pancreatic Cancer Action Network
Locations (2):
- United States (2):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - New York University, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Babb J, Rogatko A, Zacks S. Cancer phase I clinical trials: efficient dose escalation with overdose control. Stat Med. 1998 May 30;17(10):1103-20. doi: 10.1002/(sici)1097-0258(19980530)17:103.0.co;2-9. PMID 9618772
- [Background] Das S, Shapiro B, Vucic EA, Vogt S, Bar-Sagi D. Tumor Cell-Derived IL1beta Promotes Desmoplasia and Immune Suppression in Pancreatic Cancer. Cancer Res. 2020 Mar 1;80(5):1088-1101. doi: 10.1158/0008-5472.CAN-19-2080. Epub 2020 Jan 8. PMID 31915130
- [Background] FDA, Challenges and Opportunities Report. Innovation or Stagnation: Challenge and Opportunity on the Critical Path to New Medical Products. March 2004.
- [Background] Kaplanov I, Carmi Y, Kornetsky R, Shemesh A, Shurin GV, Shurin MR, Dinarello CA, Voronov E, Apte RN. Blocking IL-1beta reverses the immunosuppression in mouse breast cancer and synergizes with anti-PD-1 for tumor abrogation. Proc Natl Acad Sci U S A. 2019 Jan 22;116(4):1361-1369. doi: 10.1073/pnas.1812266115. Epub 2018 Dec 13. PMID 30545915
- [Background] Neuenschwander B, Branson M, Gsponer T. Critical aspects of the Bayesian approach to phase I cancer trials. Stat Med. 2008 Jun 15;27(13):2420-39. doi: 10.1002/sim.3230. PMID 18344187
- [Background] Neuenschwander B, Capkun-Niggli G, Branson M, Spiegelhalter DJ. Summarizing historical information on controls in clinical trials. Clin Trials. 2010 Feb;7(1):5-18. doi: 10.1177/1740774509356002. PMID 20156954
- [Background] Neuenschwander B, Wandel S, Roychoudhury S, Bailey S. Robust exchangeability designs for early phase clinical trials with multiple strata. Pharm Stat. 2016 Mar-Apr;15(2):123-34. doi: 10.1002/pst.1730. Epub 2015 Dec 18. PMID 26685103
- [Background] Nomi T, Sho M, Akahori T, Hamada K, Kubo A, Kanehiro H, Nakamura S, Enomoto K, Yagita H, Azuma M, Nakajima Y. Clinical significance and therapeutic potential of the programmed death-1 ligand/programmed death-1 pathway in human pancreatic cancer. Clin Cancer Res. 2007 Apr 1;13(7):2151-7. doi: 10.1158/1078-0432.CCR-06-2746. PMID 17404099
- [Background] Natanegara F, Neuenschwander B, Seaman JW Jr, Kinnersley N, Heilmann CR, Ohlssen D, Rochester G. The current state of Bayesian methods in medical product development: survey results and recommendations from the DIA Bayesian Scientific Working Group. Pharm Stat. 2014 Jan-Feb;13(1):3-12. doi: 10.1002/pst.1595. Epub 2013 Sep 11. PMID 24027093
- [Background] Spiegelhalter, DJ. Incorporating Bayesian Ideas into Health-Care Evaluation. Statistical Science, 2004. 19(1), 156-174.
- [Background] Von Hoff DD, Ramanathan RK, Borad MJ, Laheru DA, Smith LS, Wood TE, Korn RL, Desai N, Trieu V, Iglesias JL, Zhang H, Soon-Shiong P, Shi T, Rajeshkumar NV, Maitra A, Hidalgo M. Gemcitabine plus nab-paclitaxel is an active regimen in patients with advanced pancreatic cancer: a phase I/II trial. J Clin Oncol. 2011 Dec 1;29(34):4548-54. doi: 10.1200/JCO.2011.36.5742. Epub 2011 Oct 3. PMID 21969517

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants received 250mg s.c. Canakinumab and 400mg Spartalizumab Q4W and Gemcitabine/nab-paclitaxel per study design. No dose de-escalation occurred.
Groups:
- 250 mg s.c. Q4W Canakinumab: The study treatment is defined as spartalizumab with canakinumab in combination with gemcitabine and nab-paclitaxel.
Period: Overall Study
Arm/Group | 250 mg s.c. Q4W Canakinumab
Started | 10
Completed | 4
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | 250 mg s.c. Q4W Canakinumab
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (7.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10
Height [Mean (Standard Deviation); unit: cm] | 170.12 (8.444)
Weight [Mean (Standard Deviation); unit: kg] | 72.80 (12.251)
Body Mass Index (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 25.84 (3.688)
Baseline Body Surface Area (m^2) [Mean (Standard Deviation); unit: m^2] | 1.84 (0.174)
Childbearing potential for females [Count of Participants; unit: Participants] — Population: Count of female participants.
  Participants
    number analyzed (Participants) | 5
    Yes | 0
    No | 5

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of DLTs in the First 56 Days (8 Weeks) of Dosing to Determine Tolerable Phase 2/3 Dose of Canakinumab, Spartalizumab, Nab-paclitaxel and Gemcitabine in Patients With Metastatic Pancreatic Cancer.
Description: Evaluate dose limiting toxicities of patients with metastatic pancreatic cancer for at least 56 days (DLT period) after dosing with canakinumab at 250 mg every 4 weeks (Q4W), 400mg Spartalizumab Q4W and Gemcitabine/nab-paclitaxel on Days 1, 8 and 15 at standard of care levels. Dose limiting toxicities were evaluated to determine if dosing of canakinumab at 250 mg every 4 weeks with the other three drugs was considered tolerable and should be the dose utilized for future Phase 2/3 clinical trials. The starting dose level of canakinumab explored was 250 mg every 4 weeks (Q4W) ("starting dose level"). In case of unacceptable toxicity of canakinumab at 250 mg Q4W, the dose of canakinumab was to be de-escalated to 250 mg every 8 weeks, while other components of the combination were kept at the same dose as the starting dose level. Approximately 10 patients were to be enrolled in this study to have at least 6 evaluable patients per dose level of canakinumab.
Time Frame: Assess the incidence of dose limiting toxicities (DLT) in the first 56 days (8 weeks) of dosing
Population: Included all patients from the safety analysis set who met the minimum exposure criterion and had sufficient safety evaluations or experienced a DLT during the first 2 cycles (56 days [8 weeks]) of dosing.
Measure: Count of Participants; unit: Participants
Arm/Group | 250 mg s.c. Q4W Canakinumab
Number analyzed (Participants) | 6
Participants
  Patients with no DLTs during DLT period | 5
  Patients with DLTs including grade 4 neutropenia of Unknown duration during DLT period | 1

2. Secondary Outcome: To Determine the Safety and Tolerability of Canakinumab in Combination With Spartalizumab, Nab-paclitaxel, and Gemcitabine
Description: Determine the Safety of canakinumab, spartalizumab, nab-paclitaxel and gemcitabine via frequency and severity of adverse events (AEs), serious and non-serious. To assess tolerability of canakinumab, spartalizumab, nab-paclitaxel and gemcitabine via frequency of dose interruptions and dose reductions
Time Frame: From Day 1 of study treatment through Safety Follow-up period (150-days after the last study treatment)
Population: Included all patients treated with at least 1 dose of any of the constituent study treatments.
Measure: Number; unit: participants
Arm/Group | 250 mg s.c. Q4W Canakinumab
Number analyzed (Participants) | 10
participants
  Any TEAE | 10
  Any TEAE causally related to any drug | 10
  Any TEAE of CTCAE grade ≥3 causally related to any drug | 9
  Any TEAE with outcome of death | 0
  Any TESAE | 7
  Any TESAE causing discontinuation of any drug | 2
  Any TEAE causing discontinuation of any drug | 2
  Any TEAE leading to dose interval modified of canakinumab | 2
  Any TEAE leading to dose interruption of spartalizumab | 3
  Any TEAE leading to dose interruption of nab-paclitaxel | 7
  Any TEAE leading to dose interruption of gemcitabine | 7
  Any TEAE causing discontinuation of canakinumab causally related to any drug | 1

3. Secondary Outcome: Determine the Tolerability of Canakinumab, Spartalizumab, Nab-paclitaxel and Gemcitabine in Patients With Metastatic Pancreatic Cancer
Description: Determine the Tolerability through frequency of dose interruptions and dose reductions of canakinumab, spartalizumab, nab-paclitaxel and gemcitabine
Time Frame: From Day 1 of study treatment through End of Treatment visit, an average of 6 months
Population: Included all patients treated with at least 1 dose of any of the constituent study treatments.
Measure: Number; unit: participants
Arm/Group | 250 mg s.c. Q4W Canakinumab
Number analyzed (Participants) | 10
participants
  Number of Patients with a Reduction in Frequency from Q4W to Q8W of Canakinumab | 0
  Number of Patients with a Dose Reduction of Canakinumab | 0
  Number of Patients with neither Dose Interruption nor Dose Reduction of Spartalizumab | 10
  Number of Patients with at least one Dose Interruption or Dose Reduction of Nab-Paclitaxel | 6
  Number of Patients with at least one Dose Interruption or Dose Reduction of Gemcitabine | 6

4. Secondary Outcome: Determine the Response-related Efficacy Assessments Objective Response Rate (ORR) and Duration of Response (DOR) of Canakinumab, Spartalizumab, Nab-paclitaxel and Gemcitabine in Patients With Metastatic Pancreatic Cancer
Description: Objective Response Rate (ORR) and Duration of Response (DOR) are calculated based on tumor response data [complete Response (CR) and Partial Response (PR)] assessed at the local site using RECIST 1.1 Criteria of patients treated with canakinumab, spartalizumab, nab-paclitaxel and gemcitabine. Per Overall Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT Scans: Complete Response(CR), Disappearance of all target and non-target lesions; Partial Response (PR), at least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.; Objective/Overall Response Rate (ORR) = CR or PR.
Time Frame: Tumor response data from CT/MRI scans will be taken at screening visit and every 8 weeks throughout study treatment, an average of 6 months;
Population: Objective response rate is defined as the proportion of patients with Best Overall Response (BOR) of CR or PR per RECIST v1.1 and will be based on a subset of all treated patients with measurable disease at baseline per the site investigator.
Measure: Number; unit: participants
Arm/Group | 250 mg s.c. Q4W Canakinumab
Number analyzed (Participants) | 10
participants
  Achieved Complete Response | 0
  Achieved Partial Response | 2

5. Secondary Outcome: Determine the Disease Control Rate (DCR) of Canakinumab, Spartalizumab, Nab-paclitaxel and Gemcitabine in Patients With Metastatic Pancreatic Cancer
Description: The Disease Control Rate (DCR) is calculated based on tumor response data [complete Response (CR) and Partial Response (PR) and Stable Disease (SD)] assessed at the local site using RECIST 1.1 Criteria of patients treated with canakinumab, spartalizumab, nab-paclitaxel and gemcitabine
Time Frame: as for outcome 4
Population: DCR is defined as the proportion of patients with a BOR of CR, PR or SD (without subsequent cancer therapy) for at least 7 weeks after start of treatment as per RECIST v1.1 and will be based on a subset of all treated patients with measurable disease at baseline per the site investigator
Measure: Count of Participants; unit: Participants
Arm/Group | 250 mg s.c. Q4W Canakinumab
Number analyzed (Participants) | 10
Participants
  Disease Control | 8
  Progression | 2

6. Secondary Outcome: Determine the Progression Free Survival (PFS) of Canakinumab, Spartalizumab, Nab-paclitaxel and Gemcitabine in Patients With Metastatic Pancreatic Cancer
Description: The Progression Free Survival is defined as the time from the date of the first dose to the date of disease progression, assessed at the local site using RECIST 1.1 Criteria, of patients treated with canakinumab, spartalizumab, nab-paclitaxel and gemcitabine
Time Frame: as for outcome 4
Population: Included all patients treated with at least 1 dose of any of the constituent study treatments and both screening and on treatment study scans.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 250 mg s.c. Q4W Canakinumab
Number analyzed (Participants) | 10
months | 4.60 [1.875 to 7.566]

7. Secondary Outcome: Determine the Time To Response Rate (TTR) of Canakinumab, Spartalizumab, Nab-paclitaxel and Gemcitabine in Patients With Metastatic Pancreatic Cancer
Description: The Time To Response Rate is defined as the time from the date of the first dose to the date of first documented tumor response [Complete Response (CR) or Partial Response (PR)], assessed at the local site using RECIST 1.1 Criteria, of patients treated with canakinumab, spartalizumab, nab-paclitaxel and gemcitabine. TTR is only assessed for patients with either CR or PR.
Time Frame: as for outcome 4
Population: Included all patients treated with at least 1 dose of any of the constituent study treatments and either a CR or PR.
Measure: Median (Full Range); unit: months
Arm/Group | 250 mg s.c. Q4W Canakinumab
Number analyzed (Participants) | 2
months | 4.9 [1.71 to 8.09]

8. Secondary Outcome: Determine the Overall Survival (OS) of Canakinumab, Spartalizumab, Nab-paclitaxel and Gemcitabine in Patients With Metastatic Pancreatic Cancer
Description: The Overall Survival is defined as the time from the date of the first dose to the date of death, due to any cause, of patients treated with canakinumab, spartalizumab, nab-paclitaxel and gemcitabine
Time Frame: Overall Survival assessment will be from first day of study treatment, through safety follow up period, and until subject's date of death, or until study closure
Population: Included all patients treated with at least 1 dose of any of the constituent study treatments.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 250 mg s.c. Q4W Canakinumab
Number analyzed (Participants) | 10
months | 12.90 [3.651 to 21.711]

9. Secondary Outcome: Characterize the Pharmacokinetics of Canakinumab in Patients With Metastatic Pancreatic Cancer
Description: Characterize the Descriptive Statistics (n, m (number of non-zero concentrations), mean, coefficient of variation (CV)%, SD, median, geometric mean, geometric CV%, minimum and maximum) of the Pharmacokinetic (PK) blood samples of patients treated with canakinumab, spartalizumab, nab-paclitaxel and gemcitabine;
Time Frame: Pharmacokinetic (PK) blood draws will be taken during cycles 1-6 for canakinumab analyte; Every cycle is 28-days, total estimated time is 6 months;
Population: Pharmacokinetic analysis set (PAS) canakinumab : included all patients who received at least 1 dose of canakinumab and had at least 1 reportable concentration of canakinumab.
Measure: Median (Full Range); unit: hours (t-max)
Arm/Group | 250 mg s.c. Q4W Canakinumab
Number analyzed (Participants) | 10
hours (t-max) | 204 [142 to 506]

10. Secondary Outcome: Characterize the Pharmacokinetics of Spartalizumab in Patients With Metastatic Pancreatic Cancer
Description: Characterize the Descriptive Statistics (n, m (number of non-zero concentrations), mean, coefficient of variation CV%, SD, median, geometric mean, geometric CV%, minimum and maximum) of the Pharmacokinetic (PK) blood samples of patients treated with canakinumab, spartalizumab, nab-paclitaxel and gemcitabine;
Time Frame: Pharmacokinetic (PK) blood draws will be taken during cycles 1-6 for spartalizumab analyte; Every cycle is 28-days, total estimated time is 6 months;
Population: PAS spartalizumab : included all patients who received at least 1 dose of spartalizumab and had at least 1 reportable concentration of spartalizumab .
Measure: Median (Full Range); unit: hours (t-max)
Arm/Group | 250 mg s.c. Q4W Canakinumab
Number analyzed (Participants) | 9
hours (t-max) | 0.533 [0.500 to 0.617]

11. Secondary Outcome: Characterize the Pharmacokinetics of Nab-paclitaxel in Patients With Metastatic Pancreatic Cancer
Description: as for outcome 10
Time Frame: Pharmacokinetic (PK) blood draws will be taken during cycles 1 and 2 for nab-paclitaxel analyte; Every cycle is 28-days, total estimated time is 2 months;
Population: PAS nab-paclitaxel: included all patients who received at least 1 dose of nab-paclitaxel land had at least 1 reportable concentration of nab-paclitaxel.
Measure: Median (Full Range); unit: hours (t-max)
Arm/Group | 250 mg s.c. Q4W Canakinumab
Number analyzed (Participants) | 10
hours (t-max)
  C1D1 | 0.583 [0.567 to 0.717]
  C2D1: number analyzed (Participants) | 4
  C2D1 | 0.592 [0.533 to 0.650]

12. Secondary Outcome: Characterize the Pharmacokinetics of Gemcitabine in Patients With Metastatic Pancreatic Cancer
Description: as for outcome 10
Time Frame: Pharmacokinetic (PK) blood draws will be taken during cycles 1 and 2 for gemcitabine analyte; Every cycle is 28-days, total estimated time is 2 months;
Population: PAS gemcitabine : included all patients who received at least 1 dose of gemcitabine and had at least 1 reportable concentration of gemcitabine.
Measure: Median (Full Range); unit: hours (t-max)
Arm/Group | 250 mg s.c. Q4W Canakinumab
Number analyzed (Participants) | 10
hours (t-max)
  C1D1- GEM | 0.533 [0.400 to 0.717]
  C2D1- GEM: number analyzed (Participants) | 4
  C2D1- GEM | 0.558 [0.533 to 0.567]
  C1D1- dFdu | 0.550 [0.400 to 4.67]
  C2D1- dFdu: number analyzed (Participants) | 4
  C2D1- dFdu | 0.558 [0.533 to 0.567]

13. Other Pre Specified Outcome: Study the Immunogenicity [by Tabulating the Anti-drug Antibodies (ADA) Prevalence at Baseline and ADA Incidence On-treatment] of Canakinumab, and Spartalizumab Combined With Nab-paclitaxel and Gemcitabine in Metastatic Pancreatic Cancer Patients
Description: Study the immunogenicity [by tabulating the Anti-drug Antibodies (ADA) prevalence at baseline and ADA incidence on-treatment] of patients treated with canakinumab;
Time Frame: Immunogenicity Samples of canakinumab analytes are taken during Cycles 1-6 of study treatment; Every cycle is 28-days, total estimated time is 6 months;
Arm/Group | 250 mg s.c. Q4W Canakinumab
Number analyzed (Participants) | 0

14. Other Pre Specified Outcome: Study the Immunogenicity [by Tabulating the Anti-drug Antibodies (ADA) Prevalence at Baseline and ADA Incidence On-treatment] of Canakinumab, and Spartalizumab Combined With Nab-paclitaxel and Gemcitabine in Metastatic Pancreatic Cancer Patients
Description: Study the immunogenicity [by tabulating the Anti-drug Antibodies (ADA) prevalence at baseline and ADA incidence on-treatment] of patients treated with spartalizumab;
Time Frame: Immunogenicity Samples of spartalizumab analytes are taken during Cycles 1-6 of study treatment; Every cycle is 28-days, total estimated time is 6 months;
Arm/Group | 250 mg s.c. Q4W Canakinumab
Number analyzed (Participants) | 0

15. Other Pre Specified Outcome: Study the Immune Modulation Effect of This 4-drug Combination on the Tumor Micro-environment Using Sample Analysis From Tissue Biopsies.
Description: Study the immune modulation effect of this 4-drug combination on the tumor micro-environment from tissue biopsies, and analyzed for genomic analyses (RNA and DNA sequencing);
Time Frame: Tissue samples will be taken at two timepoints: at baseline visit (Prior to treatment) and after 8-weeks of study treatment;
Arm/Group | 250 mg s.c. Q4W Canakinumab
Number analyzed (Participants) | 0

16. Other Pre Specified Outcome: Study the Immune Modulation Effect of This 4-drug Combination on the Tumor Micro-environment Using Immunostaining From Tissue Biopsies.
Description: Study the immune modulation effect of this 4-drug combination on the tumor micro-environment from tissue biopsies, and analyzed for immunostaining;
Time Frame: as for outcome 15
Arm/Group | 250 mg s.c. Q4W Canakinumab
Number analyzed (Participants) | 0

17. Other Pre Specified Outcome: Study the Immune Modulation Effect of This 4-drug Combination on the Tumor Micro-environment Using Flow Cytometry From Tissue Biopsies.
Description: Study the immune modulation effect of this 4-drug combination on the tumor micro-environment from tissue biopsies, and analyzed for flow cytometry;
Time Frame: as for outcome 15
Arm/Group | 250 mg s.c. Q4W Canakinumab
Number analyzed (Participants) | 0

18. Other Pre Specified Outcome: Study the Immune Modulation Effect of This 4-drug Combination on the Tumor Micro-environment Using CyTOF Analysis From Tissue Biopsies.
Description: Study the immune modulation effect of this 4-drug combination on the tumor micro-environment from tissue biopsies, and analyzed for CyTOF;
Time Frame: as for outcome 15
Arm/Group | 250 mg s.c. Q4W Canakinumab
Number analyzed (Participants) | 0

19. Other Pre Specified Outcome: Study the Immune Modulation Effect of This 4-drug Combination on the Tumor Micro-environment Using Single-cell RNA Sequencing From Tissue Biopsies.
Description: Study the immune modulation effect of this 4-drug combination on the tumor micro-environment from tissue biopsies, and analyzed for single-cell RNA sequencing;
Time Frame: as for outcome 15
Arm/Group | 250 mg s.c. Q4W Canakinumab
Number analyzed (Participants) | 0

20. Other Pre Specified Outcome: To Study IL-1B Signaling by Measuring IL-6 and CRP in Serum in Human Pancreatic Ductal Adenocarcinoma (PDAC)
Description: IL-1B signaling in human PDAC will be analyzed by measuring IL-6 and CRP in serum;
Time Frame: Blood samples for these analyses will be collected during Days 1 and 15 of every treatment Cycle, on Day 8 of cycle 1, and End of Treatment Visit, an average of 6 months; ;
Arm/Group | 250 mg s.c. Q4W Canakinumab
Number analyzed (Participants) | 0

21. Other Pre Specified Outcome: To Study IL-1B Signaling by Performing ctDNA Analysis in Human Pancreatic Ductal Adenocarcinoma (PDAC)
Description: IL-1B signaling in human PDAC will be analyzed by performing ctDNA analysis;
Time Frame: as for outcome 20
Arm/Group | 250 mg s.c. Q4W Canakinumab
Number analyzed (Participants) | 0

22. Other Pre Specified Outcome: To Study IL-1B Signaling by Measuring a Panel of Cancer-related Cytokines in Plasma in Human Pancreatic Ductal Adenocarcinoma (PDAC)
Description: IL-1B signaling in human PDAC will be analyzed by measuring a panel of cancer-related cytokines in plasma;
Time Frame: as for outcome 20
Arm/Group | 250 mg s.c. Q4W Canakinumab
Number analyzed (Participants) | 0

23. Other Pre Specified Outcome: To Study IL-1B Signaling by Isolating Leukocytes in Human Pancreatic Ductal Adenocarcinoma (PDAC)
Description: IL-1B signaling in human PDAC will be analyzed by the isolation of leukocytes;
Time Frame: as for outcome 20
Arm/Group | 250 mg s.c. Q4W Canakinumab
Number analyzed (Participants) | 0

24. Other Pre Specified Outcome: To Study IL-1B Signaling by Performing Flow Cytometry in Human Pancreatic Ductal Adenocarcinoma (PDAC)
Description: IL-1B signaling in human PDAC will be analyzed by flow cytometry;
Time Frame: as for outcome 20
Arm/Group | 250 mg s.c. Q4W Canakinumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: All S/AEs, including any laboratory abnormalities, that fit the reportable criteria described in protocol, will be recorded from the time the patient signs the Informed Consent Form (ICF) until 150 days (5 months) after the last dose of study treatment of canakinumab or spartalizumab (due to the half-life of these drugs) up to 626 days/20.6 months.
Arm/Group | 250 mg s.c. Q4W Canakinumab
All-Cause Mortality (participants affected / at risk) | 9/10
Serious Adverse Events (participants affected / at risk) | 7/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 250 mg s.c. Q4W Canakinumab (N=10)
Anaemia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Gastrointestinal Disorder (Gastrointestinal disorders) | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1
Influenza Like Illness (General disorders) | 1
Biliary Obstruction (Hepatobiliary disorders) | 1
Device Related Infection (Infections and infestations) | 1
Liver Abscess (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Septic Shock (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Acute Kidney Injury (Renal and urinary disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Peripheral Ischaemia (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 250 mg s.c. Q4W Canakinumab (N=10)
Anaemia (Blood and lymphatic system disorders) | 10
Neutropenia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Sinus tachycardia (Cardiac disorders) | 1
Hypothyroidism (Endocrine disorders) | 3
Hyperthyroidism (Endocrine disorders) | 3
Retinopathy (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 6
Abdominal pain (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 4
Stomatitis (Gastrointestinal disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 8
Oedema peripheral (General disorders) | 4
Pyrexia (General disorders) | 3
Influenza like illness (General disorders) | 2
Non-cardiac chest pain (General disorders) | 2
Malaise (General disorders) | 1
Biliary obstruction (Hepatobiliary disorders) | 1
Pneumonia (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Device related infection (Infections and infestations) | 1
Liver abscess (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Vulvovaginal mycotic infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 9
Aspartate aminotransferase increased (Investigations) | 9
Blood alkaline phosphatase increased (Investigations) | 6
Neutrophil count decreased (Investigations) | 6
Platelet count decreased (Investigations) | 6
Lipase increased (Investigations) | 4
Lymphocyte count decreased (Investigations) | 4
White blood cell count decreased (Investigations) | 4
Amylase increased (Investigations) | 3
Weight decreased (Investigations) | 3
Blood bilirubin increased (Investigations) | 2
Blood creatinine increased (Investigations) | 2
Blood lactate dehydrogenase increased (Investigations) | 2
Activated partial thromboplastin time prolonged (Investigations) | 1
Blood thyroid stimulating hormone decreased (Investigations) | 1
Blood thyroid stimulating hormone increased (Investigations) | 1
International normalised ratio increased (Investigations) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6
Decreased appetite (Metabolism and nutrition disorders) | 4
Hyponatraemia (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Dysgeusia (Nervous system disorders) | 5
Peripheral sensory neuropathy (Nervous system disorders) | 3
Aphasia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 3
Anxiety (Psychiatric disorders) | 2
Pollakiuria (Renal and urinary disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2
Allergic cough (Reproductive system and breast disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1
Nail pigmentation (Skin and subcutaneous tissue disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Peripheral ischaemia (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-16): https://cdn.clinicaltrials.gov/large-docs/43/NCT04581343/Prot_SAP_000.pdf